CLINICAL TRIAL: NCT05918757
Title: Exploratory Study to Evaluate the Efficacy and Safety of Nutritional Administration of 1.5 g of Protein/kg/Day Versus 1.0 g of Protein/kg/Day in the Catabolic Phase of Critically Ill Patients Receiving Mechanical Ventilation.
Brief Title: Efficacy and Safety of Administration of High Levels of Protein to Critically Ill Patients.
Acronym: FISIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Society of Critical Care Medicine and Coronary Units (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASF1; 2021-002329-56 (EudraCT Number)
Record Dates: First submitted 2023-05-30; First posted 2023-06-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Intensive Care Unit Acquired Weakness
Keywords: Critically ill; Mechanical ventilation; Parenteral nutrition; Enteral nutrition; Protein dose
MeSH Terms: conditions — Critical Illness; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Within 48 hours, intensive care patients on expected invasive mechanical ventilation of at least three days are allocated into two groups receiving enteral/parenteral nutrition with 1.5 g of protein/kg/day or 1.0 g of protein/kg/day as an active comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein dose 1.5 g/kg/day (Experimental): Administration of 1.5 g of protein/kg/day in critically ill patients receiving invasive mechanical ventilation
  Interventions: Other: Protein dose 1.5 g/kg/day
- Protein dose 1.0 g/kg/day (Active Comparator): Administration of 1.0 g of protein/kg/day in critically ill patients receiving invasive mechanical ventilation
  Interventions: Other: Protein dose 1.0 g/kg/day

INTERVENTIONS:
Other: Protein dose 1.5 g/kg/day — Administration of 1.5 g of protein/kg/day via enteral/parenteral nutrition
  Arms: Protein dose 1.5 g/kg/day
Other: Protein dose 1.0 g/kg/day — Administration of 1.0 g of protein/kg/day via enteral/parenteral nutrition
  Arms: Protein dose 1.0 g/kg/day

SUMMARY:
Critically ill patients are known to develop serious nutritional deterioration during the course of their disease. They develop, from the beginning, a multifactorial protein malnutrition that relates to a poor clinical course and the development of weakness. Due to the increased protein catabolism in this type of patient, there is a rapid degradation of muscle mass and loss of functional proteins, and therefore nutritional support is mandatory. Indeed, achieving a high protein intake may promote a better evolution of the critically ill patient, i.e., maintenance of muscle protein, less deterioration of muscle strength, lower Intensive care unit-acquired weakness (ICUAW), lower mortality, decrease in the number of infections, decrease in days on mechanical ventilation, and days of hospital stay and in ICU.

The goal of this clinical trial is to compare the appearance and degree of ICUAW in critically ill patients receiving invasive mechanical ventilation treated with two different doses of protein (1.5 g/kg/day vs.1.0 g/kg/day).

DETAILED DESCRIPTION:
It is known that protein metabolism is altered in critically ill patients due to metabolic alterations derived from stress. This critical situation is manifested by a severe catabolic alteration, especially in the first week, which is fundamentally characterized by severe glucose intolerance and the use of the protein itself as a metabolic substrate.

Despite protein synthesis is increased, this is insufficient to compensate for the high protein degradation rate, which leads, among others, to muscle deterioration resulting in increased morbidity and mortality. This muscle destruction has been implicated in the early appearance of Intensive care unit-acquired weakness (ICUAW). Although the pathophysiology of ICUAW is multifactorial, protein intake may play an key role in its treatment. However, protein intake cannot reduce muscle destruction, but it can stimulate protein synthesis.

Current evidence supports that the administration of early artificial nutritional support with a high protein intake can improve the clinical course of critically ill patients. However, there is still no consensus on the exact amount of protein needed to be administered to these patients in order to reduce adverse outcomes and prevent ICUAW.

Thus the aim of this study is to evaluate the effect of a nutritional supplementation containing 1.5 g of protein/kg/day vs 1.0 g of protein /kg/day in critically ill patients receiving mechanical ventilation on the development and degree of ICUAW.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patient
* ICU admission during the previous 48h
* Patients on expected invasive mechanical ventilation for three days
* Patients with a minimum expected duration of clinical nutrition of at least seven days
* Written informed consent signed by the patient or the patient's legally authorized representative.
* Available central venous access for continuous infusion of the study drugs.

Exclusion Criteria:

* Denied informed consent
* Acute renal failure (renal injury stage 3)
* Liver failure (cirrhosis or Child-Pugh Scale > 5)
* Severe liver failure with International Normalized Ratio (INR) > 1.7 (prothrombin time > 50%) and encephalopathy
* Patients with COVID-19-derived pneumonia
* Body Mass Index (BMI) > 40 or < 18.5 (morbid obesity or previous caloric malnutrition)
* Pregnant patients
* Central Nervous System pathologies (Glasgow < 6)
* Peripheral Nervous System pathologies interfering with study evaluations
* Patients with cognitive dysfunction/dementia or unable to follow instructions regarding MRC tests
* Severe muscular pathology
* Already participating in another clinical trial
* Impossibility to contact after ICU discharge to carry out the follow-up visit on day 90
* Known hypersensitivity to milk protein or any of the components of the nutritional supplement
* Inborn errors in the amino acid metabolism
* Previous inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of intensive care unit acquired weakness (ICUAW). | Baseline, weekly in ICU up to 28 days after mechanical ventilation termination, throughout hospital stay, an expected average of 6 weeks, and 90 days after hospital discharge.
  Determined by Medical Research Council sum score (MRC-SS). Diagnosis of ICUAW if MRC-SS < 48 (maximun score 60).

SECONDARY OUTCOMES:
Muscle Strength. | Up to 6 months.
  Dynamometry.
Active mobility. | Up to 6 months.
  Determined by Intensive Care Unit Mobility Scale (ICUMS). Scored from 0 to 10 being 0 no activity, lying in bed, and 10 walking independently without a gait aid.
Nosocomial infections. | Throughout hospital stay, an expected average of 6 weeks.
  Centers for disease control and prevention (CDC).
Mechanical ventilation. | Up to 1 month.
  Number of days receiving mechanical ventilation.
Gastrointestinal complications. | Throughout hospital stay, an expected average of 6 weeks.
  Gastric residual volume, diarrhea, vomiting or regurgitation, abdominal distension, constipation.
Metabolic complications. | Throughout hospital stay, an expected average of 6 weeks.
  Glycemia, fluid intake, electrolytes/trace element determination, hypertriglyceridemia, liver disfunction, cholestasis, necrosis or mixed dysfunction, overfeeding.
Mortality rate. | Up to 6 months.
  Number of deaths/total participants
Length of ICU and hospital stay. | Throughout hospital stay, an expected average of 6 weeks.
  Number of days of hospitalization.
Quality of life index. | Up to 6 months.
  European Quality of Life-5 Dimensions (EQ-5D). Scored from 0 to 100 being 0 the worst health imaginable and 100 the best health imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: María Carmen Sánchez Álvarez, PhD, Principal Investigator — Sociedad Española de Medicina Intensiva, Crítica y Unidades Coronarias (SEMICYUC); Juan Francisco Fernández Ortega, PhD, Principal Investigator — Hospital Regional de Malaga
Locations (18):
- Spain (18):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario de Castellón, Castellon, Castelló
  - Hospital Universitario de Badajoz, Badajoz, Extremadura
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital de Manacor, Manacor, Mallorca
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital General Universitario Los Arcos del Mar Menor, Pozo-Aledo, Murcia
  - Hospital Universitario Doctor Josep Trueta, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario San Jorge, Huesca
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia

IPD SHARING:
Plan to Share IPD: No